CLINICAL TRIAL: NCT04666311
Title: Prospective, Multicentre Evaluation of the Accuracy of CAD4TB and C-reactive Protein Assay as Triage Tests for the Diagnosis of Pulmonary Tuberculosis in Presumptive Adult TB Patients (TB TRIAGE+ Accuracy)
Brief Title: Diagnostic Accuracy of CAD4TB and C-reactive Protein Assay as Triage Tests for Pulmonary Tuberculosis
Acronym: TB TRIAGE+
Status: Completed | Type: Observational
Sponsor: Klaus Reither (Other)
Collaborators: SolidarMed (Other); Human Sciences Research Council (Other Government); Institute of Tropical Medicine, Belgium (Other); Radboud University Medical Center (Other); Charite University, Berlin, Germany (Other); University Hospital, Basel, Switzerland (Other); Foundation for Innovative New Diagnostics, Switzerland (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Ministry of Health, Lesotho (Other Government)
Responsible Party: Sponsor-Investigator, Klaus Reither, Head of Clinical Research Unit, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Other Study IDs: P1685-20A
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Tuberculosis; Tuberculosis Diagnosis; Covid-19; HIV
Keywords: Presumptive adult TB; C Reactive Protein assay; CAD4TB; Point of Care Test; TB Triage Test; Diagnostic Accuracy; CAD4COVID; COVID-19 RDT; Advanced HIV Disease (AHD) care package; HIV testing; Community-based triage testing for TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; COVID-19; Alagille Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult presumptive TB cases: Adult presumptive TB cases (age ≥18years) with one or more TB symptoms (WHO recommended four-symptom screening; cough, weight loss, night sweats, fever) of any duration.
  Interventions: Diagnostic Test: Accuracy of CAD4TB and Afinion CRP assay for pulmonary TB; Diagnostic Test: CAD4COVID+WBC and COVID-19 RDT for SARS-CoV-2 infection

INTERVENTIONS:
Diagnostic Test: Accuracy of CAD4TB and Afinion CRP assay for pulmonary TB — CAD4TB version 6 and 7: Software tool for detecting lung abnormalities in computer tomogram images (pulmonary abnormalities) and frontal chest radiograph images (tuberculosis abnormalities) ; availability is guaranteed by Delft Imaging System; EC 0344 Certificate (vs.6); CE mark pending (vs.7). Will be performed by a registered and qualified radiographer in accordance with national regulations.
  Afinion AS100 Analyzer and Afinion CRP: In vitro diagnostic to determine the amount of CRP in human whole blood, serum or plasma; CE-mark ; Will be performed by qualified, GCP-trained study personnel.
Diagnostic Test: CAD4COVID+WBC and COVID-19 RDT for SARS-CoV-2 infection — CAD4COVID: Non-commercial product. Software tool for detecting pneumonia-related features to be expected in COVID-19 patients; availability is guaranteed by Delft Imaging System; CE certified. Will be performed by a registered and qualified radiographer/health professional in accordance with national regulations. Analysis in combination with differential white blood cell count.
  SD Biosensor, STANDARDTM Q COVID-19 Ag Test (rapid chromatographic immunoassay for the qualitative detection of specific antigens to SARS-CoV-2)

SUMMARY:
In the TB TRIAGE+ ACCURACY study, the accuracy of the following products will be determined:

* CAD4TB (Delft Imaging System, NL), a digital chest x-ray analysis software
* Afinion CRP assay (Alere Afinion, USA), which detects a cytokine induced acute phase protein

CAD4TB and the C-reactive protein assay are two tests with great potential of becoming a triage test for the diagnosis of tuberculosis (TB). These potential triage tests for TB are intended to serve as rule-out tests with a high sensitivity and negative predictive value.

Before impact and cost-effectiveness of new TB triage tests for intensified active case finding can be determined, the diagnostic test accuracy needs to be assessed in comparison to confirmatory reference tests. This accuracy study will define cut-off values for CAD4TB as well as for the Afinion CRP assay to be used in a future cluster-randomised trial on impact and cost-effectiveness of TB triage strategies for intensified active case finding in Lesotho and KwaZulu-Natal, South Africa.

A sub-study (detailed in a separate study protocol), hereafter called AHD-FEASIBILITY, explores the feasibility of implementing a series of point-of-care tests, including the new VISITECT CD4 Advanced Disease Test (Omega Diagnostics, UK) as part of the WHO-recommended advanced HIV Disease care package in the context of community-based HIV/TB campaigns.

Due to the coinciding pandemics and the overlapping symptoms of TB and COVID-19, it is critical to test for SARS-Cov-2 infections in the study population. In addition, this study will contribute to the evaluation of a novel SARS-Cov-2 antigen rapid diagnostic test (from the diagnostic pipeline of FIND) and CAD4COVID, a digital chest x-ray analysis software (Delft Imaging System, NL) in combination with differential white blood cell count.

DETAILED DESCRIPTION:
This is a prospective, partially blinded, two-centre cross-sectional study in which the diagnostic test accuracy of CAD4TB and an Afinion CRP assay test for TB will be assessed at facility level by evaluating a sample of 1400 adults (age ≥18years) with one or more TB symptoms (WHO recommended four-symptom screening; cough, weight loss, night sweats, fever) of any duration.

Presumptive TB patients will be recruited (i) at the outpatient departments of the Butha-Buthe District Hospital (Butha-Buthe, Lesotho) and the Caluza Clinic (Pietermaritzburg, KwaZulu-Natal, South Africa) and (ii) during community-based health campaigns by SolidarMed in Lesotho and HSRC in South Africa. Participants will be enrolled after giving written informed consent.

Study procedures comprise the following (detailed in the schedule of events): collection of contact, anthropometric, demographic and clinical data, HIV testing and counselling per national guidelines, collection of capillary blood for HIV testing, Afinion CRP assay, differential white blood cell count, VISITECT CD4 Advanced Disease Test (if HIV-positive), CrAg Lateral Flow Assay (if HIV positive and CD4 count <200 cells/μl as per VISITECT CD4 Advanced Disease Test, and no history of cryptococcal meningitis treatment); collection of urine (if HIV positive) for Alere Determine TB LAM Ag test; chest radiography for CAD4TB and CAD4COVID analysis and remote expert reading; nasopharyngeal swabs for SARS-Cov-2 real-time PCR and SARS-Cov-2 antigen test, collection of two spot sputa samples (S1,S2) for Xpert MTB/RIF, Xpert MTB/RIF Ultra (S1) and for mycobacterial culture [MGIT] (S2). At week 12 (±2weeks), we will contact each participant by phone and collect data on their vital status, and any TB treatment since enrolment. For individuals on TB treatment, further information, e.g. on reasons for empirical treatment, will be collected at the health facility the participant started TB treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed written consent or witnessed oral consent in the case of illiteracy, prior to undertaking any study-related procedure
2. Adults (≥18 years)
3. Any of the cardinal symptoms of TB (cough, weight loss, night sweats, fever) of any duration

Exclusion Criteria:

1. Pregnancy (based on oral information from participant)
2. Any condition for which participation in the study, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments
3. Critically sick patients who need immediate medical care
4. Current anti-TB treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult presumptive TB cases (age ≥18years) with one or more TB symptoms (WHO recommended four-symptom screening; cough, weight loss, night sweats, fever) of any duration.
  Presumptive TB patients will be recruited (i) at the outpatient departments of the Butha-Buthe District Hospital (Butha-Buthe, Lesotho) and the Caluza Clinic (Pietermaritzburg, KwaZulu-Natal, South Africa) and (ii) during community-based health campaigns by SolidarMed in Lesotho and HSRC in South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Determine CAD4TB cut-off value | 15 months after first patient visit
  Receiver operating characteristic analysis (ROC) of CAD4TB against a composite microbiological reference standard (mycobacterial culture [MGIT] or Xpert MTB/RIF) to define an acceptable diagnostic cut-off value.
Determine Afinion CRP assay cut-off value | 15 months after first patient visit
  Receiver operating characteristic analysis (ROC) of Afinion CRP assay against a composite microbiological reference standard (mycobacterial culture [MGIT] or Xpert MTB/RIF) to define an acceptable diagnostic cut-off value.

SECONDARY OUTCOMES:
Evaluate CAD4TB ROC against reference standard | 15 months after first patient visit
  Receiver operating characteristic analysis (ROC) of CAD4TB against a single microbiological reference standard (mycobacterial culture [MGIT] alone, Xpert MTB/RIF alone, Xpert MTB/RIF Ultra alone), against a composite reference standard and against a radiological reference standard
Evaluate Afinion CRP assay ROC against reference standard | 15 months after first patient visit
  Receiver operating characteristic analysis (ROC) of Afinion CRP assay against a single microbiological reference standard (mycobacterial culture [MGIT] alone, Xpert MTB/RIF alone, Xpert MTB/RIF Ultra alone) and against a composite reference standard
Evaluate CAD4COVID and COVID-19 RDT ROC against reference standard | 15 months after first patient visit
  Receiver operating characteristic analysis (ROC) of CAD4COVID combined with differential white blood cell count and point estimates of sensitivity and specificity the novel SARS-Cov-2 antigen rapid diagnostic test, both against a single microbiological reference standard (SARS-Cov-2 real-time PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Reither, MD, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (2):
- Butha-Buthe District Hospital, Butha-Buthe, Lesotho
- Caluza Clinic, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All data will be stored securely in a way that allows future access for the research team. We will adhere to the FAIR Guiding Principles for data management and stewardship 20. After completion of the studies and after anonymization (e.g. replace subject identifier with a new random subject identifier), analysis datasets will be made publicly available in a timely manner on a non-commercial data platform according to the FAIR principles. The principles of data sharing will be explained in the informed consent form. All data will be owned by the Sponsor-Investigator and investigators of TB TRIAGE+, while a Data Access Committee will review all requests for data sharing.
Time Frame: 12 months after completion of the EDCTP-funded TB TRIAGE+ project
Access Criteria: The Executive Group of the TB TRIAGE+ project will establish a Data Access Committee (DAC). The DAC will review all requests for data sharing. After approval by the DAC, the final verified and anonymised datasets and support for analysis will be made available to all relevant stakeholders, both at local level (health facility, region and country) as well as international decision makers (e.g. WHO) and interested research groups in order to advance research in TB.

REFERENCES:
- [Result] Glaser N, Bosman S, Madonsela T, van Heerden A, Mashaete K, Katende B, Ayakaka I, Murphy K, Signorell A, Lynen L, Bremerich J, Reither K. Incidental radiological findings during clinical tuberculosis screening in Lesotho and South Africa: a case series. J Med Case Rep. 2023 Aug 25;17(1):365. doi: 10.1186/s13256-023-04097-4. PMID 37620921
- [Result] Bosman S, Ayakaka I, Muhairwe J, Kamele M, van Heerden A, Madonsela T, Labhardt ND, Sommer G, Bremerich J, Zoller T, Murphy K, van Ginneken B, Keter AK, Jacobs BKM, Bresser M, Signorell A, Glass TR, Lynen L, Reither K. Evaluation of C-Reactive Protein and Computer-Aided Analysis of Chest X-rays as Tuberculosis Triage Tests at Health Facilities in Lesotho and South Africa. Clin Infect Dis. 2024 Nov 22;79(5):1293-1302. doi: 10.1093/cid/ciae378. PMID 39190813
- [Derived] Gils T, Lynen L, Muhairwe J, Mashaete K, Lejone TI, Joseph P, Ngubane T, Keter AK, Reither K, van Heerden A. Feasibility of implementing the advanced HIV disease care package as part of community-based HIV/TB activities: a mixed-methods study protocol. BMJ Open. 2022 Feb 7;12(2):e057291. doi: 10.1136/bmjopen-2021-057291. PMID 35131835